CLINICAL TRIAL: NCT00727649
Title: Efficacy and Mechanisms of Pharmacologic Treatment of Fecal Incontinence
Acronym: FIRM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B6126-W
Record Dates: First submitted 2008-07-29; First posted 2008-08-04 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; adults; diarrhea
MeSH Terms: conditions — Fecal Incontinence; Diarrhea | interventions — Psyllium; Loperamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Fiber (psyllium) powder
  Interventions: Drug: Psyllium powder
- Arm 2 (Active Comparator): Loperamide
  Interventions: Drug: Loperamide

INTERVENTIONS:
Drug: Psyllium powder — 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose)
  Other Names: Metamucil
  Arms: Arm 1
Drug: Loperamide — 1 capsule daily for 28 days (weekly adjusted dose)
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate and compare treatment with fiber and loperamide for fecal incontinence.

DETAILED DESCRIPTION:
Fecal incontinence (FI) affects 4-24% adults in the community and greatly impacts quality of life. Both fiber and loperamide are common, first-line treatments for diarrhea-associated FI in primary care. No known studies exist that compare fiber and loperamide for diarrhea-predominant FI. Further knowledge is needed to define which treatment is more effective and to compare drug tolerability (side effects) for FI. This study will also look at changes in quality of life with treatment and potential mechanisms of drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* weekly fecal incontinence

Exclusion Criteria:

* fecal impaction
* inability to complete a baseline 1-week bowel diary
* rectal prolapse
* any prior radiation to the pelvis
* colo-rectal cancer
* rectal fistula
* inflammatory bowel disease
* neurological diseases (spinal cord injury, multiple sclerosis, Parkinson's disease)
* constipation (<2 bowel movements/week) or total colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alayne D Markland, DO MSc, Principal Investigator — VA Medical Center, Birmingham
Locations (1):
- VA Medical Center, Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient medical clinic
Groups:
- P1L2 (Psyllium First, Then Loperamide): Fiber (psyllium) powder with loperamide placebo first
  Psyllium powder: 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose) Loperamide placebo: 1 tablet daily with weekly dose adjustments for side-effects and/or efficacy
- L1P2 (Loperamide First, Then Pysllium): Fiber (psyllium) powder placebo with loperamide 2mg
  Psyllium placebo powder: 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose for side-effects and/or efficacy) Loperamide: 2 mg daily with weekly dose adjustments for side-effects and/or efficacy
Period: First Intervention (4-weeks)
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium)
Started | 37 | 43
Completed | 34 | 40
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Period: Wash-out (2-weeks)
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium)
Started | 34 | 40
Completed | 30 | 37
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2
Period: Second Intervention (4-weeks)
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium)
Started | 30 | 37
Completed | 29 | 34
Not Completed | 1 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- P1L2 (Psyllium First, Then Loperamide): Fiber (psyllium) powder with loperamide placebo first
  Psyllium powder: 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose) Loperamide placebo: 2 mg placebo daily with weekly dose adjustments for side-effects and/or efficacy
- L1P2 (Loperamide First, Then Pysllium): Fiber (psyllium) powder placebo with loperamide 2mg pill
  Psyllium placebo powder: 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose for side-effects and/or efficacy) Loperamide: 2 mg daily with weekly dose adjustments for side-effects and/or efficacy
- Total: Total of all reporting groups
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium) | Total
Number analyzed (Participants) | 37 | 43 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 33
  >=65 years | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.9) | 59.2 (9.2) | 60.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 25 | 29 | 54
Region of Enrollment [Number; unit: participants]
  United States | 37 | 43 | 80

OUTCOME MEASURES:

1. Primary Outcome: 7-day Bowel Diary, Number of Fecal Incontinence Episodes
Description: After consent, 7-day bowel diary was assessed at baseline (2-week visit), during the last week of the 4-week intervention (6-week visit), during the second week of the 2-week wash-out period at 8-weeks, and during the last week of the second 4-week intervention (12 weeks). The mean number of total fecal incontinence episodes from a 7-day bowel diary from each time point was compared between the groups.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: Fecal incontinence episodes
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium)
Number analyzed (Participants) | 34 | 39
Fecal incontinence episodes
  Baseline | 7.3 (6.2) | 7.9 (7.5)
  End of First Intervention | 4.8 (4.8) | 4.1 (5.1)
  End of Wash-out Period | 4.3 (4.2) | 5.0 (6.2)
  End of Second Intervention | 3.5 (6.6) | 4.7 (5.7)

2. Primary Outcome: Percentage of Bowel Movements With Incontinence
Description: After consent, 7-day bowel diary was assessed at baseline (2-week visit), during the last week of the 4-week intervention (6-week visit), during the second week of the 2-week wash-out period at 8-weeks, and during the last week of the second 4-week intervention (12 weeks). We compared the percentage of the total number of fecal incontinence episodes over the total number of bowel movements from a 7-day bowel diary from each time point between the groups.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of incontinent bowel movement
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium)
Number analyzed (Participants) | 34 | 39
percentage of incontinent bowel movement
  Baseline | 30.5 (18.0) | 32.3 (23.4)
  End of First Intervention | 23.4 (22.1) | 21.3 (22.7)
  End of Wash-out Period | 23.0 (22.2) | 18.8 (20.2)
  End of Second Intervention | 15.9 (19.3) | 18.8 (21.0)

3. Secondary Outcome: Fecal Incontinence Severity Index Score, FISI
Description: The patient-reported symptoms severity score, the Fecal Incontinence Severity Index (FISI), has 4 questions about the frequency of gas, mucus, liquid stool, and solid stool incontinence. Responses are weighted based on the patient rating of severity and a total score is calculated (range 0-61) with higher scores indicating a greater severity of symptoms.
Time Frame: baseline, 4 week and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | P1L2 (Psyllium First, Then Loperamide) | L1P2 (Loperamide First, Then Pysllium)
Number analyzed (Participants) | 36 | 42
units on a scale
  Baseline | 29.1 (11.0) | 31.9 (13.5)
  End of First Intervention | 24.9 (12.2) | 24.9 (13.3)
  End of Second Intervention | 22.0 (17.1) | 23.2 (12.7)

ADVERSE EVENTS:
Time Frame: We collected adverse event data during each 4-week intervention period.
Description: Weekly phone calls were made to assess symptoms and adjust medication dosages.
Groups:
- P1L2 (Psyllium First); 1st 4-weeks; L1P2 (Psyllium Second); 2nd 4-weeks: Fiber (psyllium) powder with loperamide placebo first
  Psyllium powder: 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose) Loperamide placebo: 1 tablet daily with weekly dose adjustments for side-effects and/or efficacy
- L1P2 (Loperamide First): 1st 4-weeks; P1L2 (Loperamide Second); 2nd 4-weeks: Fiber (psyllium) powder placebo with loperamide 2mg
  Psyllium placebo powder: 2 teaspoons with 8 ounces of liquid daily for 28 days (weekly adjusted dose for side-effects and/or efficacy) Loperamide: 2 mg daily with weekly dose adjustments for side-effects and/or efficacy
Arm/Group | P1L2 (Psyllium First); 1st 4-weeks | L1P2 (Loperamide First): 1st 4-weeks | P1L2 (Loperamide Second); 2nd 4-weeks | L1P2 (Psyllium Second); 2nd 4-weeks
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/40 | 1/29 | 0/34
Other Adverse Events (participants affected / at risk) | 4/34 | 6/40 | 3/29 | 4/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1L2 (Psyllium First); 1st 4-weeks (N=34) | L1P2 (Loperamide First): 1st 4-weeks (N=40) | P1L2 (Loperamide Second); 2nd 4-weeks (N=29) | L1P2 (Psyllium Second); 2nd 4-weeks (N=34)
death (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — sigmoid colon perforation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1L2 (Psyllium First); 1st 4-weeks (N=34) | L1P2 (Loperamide First): 1st 4-weeks (N=40) | P1L2 (Loperamide Second); 2nd 4-weeks (N=29) | L1P2 (Psyllium Second); 2nd 4-weeks (N=34)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (6) | 3 (3) | 2 (2)
constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3) | 3 (3)
diarrhea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 4 (4)
excessive flatus (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (3) | 4 (4)
bloating (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
heartburn (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Please note that the data on those lost to follow-up limits our ability to conclude differences between the two interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes